CLINICAL TRIAL: NCT03463837
Title: A Randomized, Open-Label, Parallel-Group Study to Characterize Biomarkers of Tobacco Exposure and Nicotine Uptake From JUUL 5% Electronic Nicotine Delivery Systems (ENDS) in Adult Smokers
Brief Title: Identify Biomarkers of Tobacco Exposure and Nicotine Uptake From JUUL 5% in Adult Smokers
Acronym: Diamond
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 755-00041
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2019-01

CONDITIONS: Nicotine Dependence, Other Tobacco Product; Tobacco Use; Smoking, Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Tobacco Smoking | interventions — Therapeutics; Mangifera indica extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment with JUUL 5%, Virginia Tobacco (Experimental): JUUL 5%,Virginia Tobacco [5 days] in confinement.
  Interventions: Other: Treatment with JUUL 5%, Virginia Tobacco
- Treatment with JUUL 5%, Cool Mint, ENDS (Experimental): JUUL 5%, Cool Mint [5 days] in confinement.
  Interventions: Other: Treatment with JUUL 5%, Cool Mint, ENDS
- Treatment with JUUL 5%, Mango, ENDS (Experimental): JUUL 5%, Mango [5 days] in confinement.
  Interventions: Other: Treatment with JUUL 5%, Mango, ENDS
- JUUL 5%, Creme Bruele, ENDS (Experimental): JUUL 5%, Creme Bruele [5 days] in confinement.
  Interventions: Other: JUUL 5%, Creme Bruele, ENDS
- Combustible cigarette (Active Comparator): Exclusive use of combustible cigarette [5 days] in confinement.
  Interventions: Other: Combustible cigarette
- Smoking cessation (no smoking) (Sham Comparator): Smoking cessation (no smoking).
  Interventions: Other: Smoking Cessation

INTERVENTIONS:
Other: Treatment with JUUL 5%, Virginia Tobacco — JUUL 5%, ENDS for 5-days in confinement
  Other Names: JUUL
  Arms: Treatment with JUUL 5%, Virginia Tobacco
Other: Treatment with JUUL 5%, Cool Mint, ENDS — JUUL 5%, ENDS for 5-days in confinement
  Other Names: JUUL
  Arms: Treatment with JUUL 5%, Cool Mint, ENDS
Other: Treatment with JUUL 5%, Mango, ENDS — JUUL 5%, ENDS for 5-days in confinement
  Other Names: JUUL
  Arms: Treatment with JUUL 5%, Mango, ENDS
Other: JUUL 5%, Creme Bruele, ENDS — JUUL 5%, ENDS for 5-days in confinement
  Other Names: JUUL
  Arms: JUUL 5%, Creme Bruele, ENDS
Other: Combustible cigarette — Exclusive use of combustible cigarette for 5 days in confinement.
  Arms: Combustible cigarette
Other: Smoking Cessation — No smoking for 5-days in confinement.
  Arms: Smoking cessation (no smoking)

SUMMARY:
The JUUL 5% Electronic Nicotine Delivery System (ENDS) is being studied as an alternative to combustible cigarette use. This study aims to find out how much nicotine is in the blood and urine of healthy adult subjects after using three JUUL 5% ENDS compared to smoking usual brands of combustible cigarettes and stopping smoking.

DETAILED DESCRIPTION:
This study will serve as a clinical evaluation of the exclusive use of selected JUUL ENDS, with the purpose of gaining an understanding of toxicant exposure.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy, adult, male or female smoker, 21 to 65 years of age.
2. Has been a smoker for at least 12 months prior to Screening.
3. Currently smokes an average of 10 cigarettes each day.
4. Has a positive urine cotinine (≥ 500 ng/mL).
5. Has an exhaled carbon monoxide (CO) > 12 ppm.
6. A female subject of childbearing potential must have been using contraception and agree to continue using it through completion of the study:
7. Provides voluntary consent to participate in this study documented on the signed informed consent form (ICF).

Key Exclusion Criteria

1. Has a history or presence of clinically significant conditions.
2. Has a body mass index (BMI) > 40 kg/m2 or < 18 kg/m2 at Screen
3. Has a history of drug or alcohol abuse
4. Has an estimated creatinine clearance < 80 mL/minute
5. If female, the subject is pregnant, lactating, or intends to become pregnant during the time period from Screening through the end of study.
6. Has used nicotine-containing products other than manufactured cigarettes within 14days of screening.
7. Is planning to quit smoking during the study, planning to quit within 3 months following Day 1

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Change in primary biomarkers day 5 values for each JUUL 5% product will be compared to baseline: | [Time Frame: 5 days]
  Change in ; Urine N nitrosonornicotine (NNN), 4 (methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), 3 hydroxypropylmercapturic acid (3-HPMA), monohydroxybutenylmercapturic acid (MHBMA), and S-phenyl mercapturic acid (S-PMA) "Blood carboxyhemoglobin (COHb)

SECONDARY OUTCOMES:
Change in concentration of 3-hydroxy-1-methylpropylmercapturic acid (HMPMA) in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of 2-cyanoethyl-mercapturic acid (CEMA) in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of 1-hydroxypyrene (1-OHP) in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of Nicotine in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of Cotinine in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of trans-3'-hydroxycotinine in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of Glucuronides in urine | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of Nicotine in blood | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of Cotinine in blood | [Time Frame: 5 days]
  Change in Biomarker
Change in concentration of trans-3'-hydroxycotinine in blood | [Time Frame: 5 days
  Change in Biomarker
Change in maximum concentration (Cmax) Plasma pharmacokinetic (PK) of Nicotine | [Time Frame: Day 7,
  Nicotine absorption
Change in time to maximum concentration (Tmax) Plasma PK of Nicotine | [Time Frame: Day 7,
  Nicotine absorption
Change of area under the curve (AUC) Plasma PK of Nicotine | [Time Frame: Day 7,
  Nicotine absorption
Product use over 5-day period and during 5-minute fixed and ad libitum use episodes | [Time Frame: 7 days]
  Change in product use
Measure of subjective Smoking Urge Assessment | [Time Frame: 6-7 days, intervention dependent]
  Change in Assessment
Measure of subjective product evaluation using the "modified Product Evaluation Scale (mPES)" | [Time Frame: 6-7 days, intervention dependent]
  Change in Evaluation; Scale: 1 = not at all, 2 = very little, 3 = a little, 4 = moderately, 5 = a lot, 6 = quite a lot, 7 = extremely
  Four multi-item subscales will be derived from "Satisfaction" (items 1, 2, 3, and 12); "Psychological Reward" (items 4 through 8); "Aversion" (items 9, 10, 16, and 18); and "Relief" (item 11, 13, 14, 15, and reversed for item 19) and single items 17 and 20 will be summarized.
Measure of future intent to use JUUL 5% Device device relative to usual combustible cigarette and smoking cessation. | [Time Frame: 6-7 days, intervention dependent]
  Change in Intent
Number of participants with Adverse Events associated with use of JUUL 5% Device to combustible cigarette and smoking cessation | [Time Frame: 13-14 days, intervention dependent]
  Safety
Incidence of JUUL 5% Device, including malfunction and/or misuse | [Time Frame: 7 days]
  Device performance

CONTACTS AND LOCATIONS:
Overall Officials: Philip Mathew, M.D., Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HIPAA Privacy Rule. Information for Researchers. De-identifying Protected Health Information Under the Privacy Rule. U.S. Department of Health and Human Services. NIH (Feb 2007). Available at: http://privacyruleandresearch.nih.gov/pr_08.asp#8a. Last accessed 31-Jul-2017.
- [Result] D'Ruiz CD, Graff DW, Robinson E. Reductions in biomarkers of exposure, impacts on smoking urge and assessment of product use and tolerability in adult smokers following partial or complete substitution of cigarettes with electronic cigarettes. BMC Public Health. 2016 Jul 11;16:543. doi: 10.1186/s12889-016-3236-1. PMID 27401980
- [Result] Jensen RP, Luo W, Pankow JF, Strongin RM, Peyton DH. Hidden formaldehyde in e-cigarette aerosols. N Engl J Med. 2015 Jan 22;372(4):392-4. doi: 10.1056/NEJMc1413069. No abstract available. PMID 25607446
- [Result] McNeill A et al. E-cigarettes: An Evidence Update. A report commissioned by Public Health England. Available at: https://www.gov.uk/government/uploads/system/uploads/ attachment_data/file/457102/Ecigarettes_an_evidence_update_A_report_commissioned_by_ Public_Health_England_FINAL.pdf (Aug 2015).
- [Result] Polosa R, Morjaria J, Caponnetto P, Caruso M, Strano S, Battaglia E, Russo C. Effect of smoking abstinence and reduction in asthmatic smokers switching to electronic cigarettes: evidence for harm reversal. Int J Environ Res Public Health. 2014 May 8;11(5):4965-77. doi: 10.3390/ijerph110504965. PMID 24814944